CLINICAL TRIAL: NCT06440070
Title: B-ultrasound-guided Bending Needle and Thread Loop Carpal Tunnel Ligament Release in Carpal Tunnel Syndrome :Efficacy and Safety of a Single-Center, Single-Arm Clinical Trial
Brief Title: Ultrasound-Guided Curved Needle Thread Carpal Tunnel Release: Efficacy and Safety of a Single-Center, Single-Arm Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-287-02
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Surgery; Ultralsound-Guide
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loop Carpal Tunnel Release group (Experimental)
  Interventions: Procedure: Loop Carpal Tunnel Release

INTERVENTIONS:
Procedure: Loop Carpal Tunnel Release — Under the guidance of ultrasound, needles are inserted above and below the transverse carpal ligament, respectively, to form a loop around the ligament. Finally, the ligament is cut by pulling the looped thread.

SUMMARY:
Carpal tunnel syndrome is a set of symptoms and signs caused by compression of the median nerve within the carpal tunnel. The prevalence in the general population is about 3.72%, with a rising trend, making it the most common peripheral nerve entrapment syndrome. Compared to conservative treatment, surgical treatment has definite efficacy and lower recurrence rates, making it the ultimate choice for relieving median nerve compression. However, open surgery has disadvantages such as large trauma, long postoperative recovery period, and scar formation, while wrist arthroscopic surgery, although minimally invasive, is technically challenging, requires expensive specialized equipment, and has low cost-effectiveness, limiting its clinical application.

Therefore, based on clinical and life experience, our team innovatively developed the "Ultrasound-guided Needle Release of the Transverse Carpal Ligament." This technique avoids the risks of large trauma and scar formation associated with traditional open surgery, significantly shortens surgical and postoperative recovery times, and is more minimally invasive and cost-effective compared to wrist arthroscopic surgery, thus having high clinical value for promotion. This study aims to validate the effectiveness and safety of this innovative procedure through a single-arm interventional clinical study, providing a theoretical basis for further clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40 and 70 years;
2. Exhibiting symptoms consistent with carpal tunnel syndrome (e.g., finger numbness, tingling, weakness, or pain; symptoms aggravated by repetitive or sustained gripping; symptoms worsening at night) and signs (sensory impairment or weakness in the hand; positive Tinel's sign or Phalen's test for the median nerve);
3. Meeting the diagnostic criteria for typical or possible carpal tunnel syndrome based on the Katz hand diagram for carpal tunnel syndrome [14];
4. Ultrasound indicating thickening of the transverse carpal ligament, compressing the median nerve;
5. Ineffective conservative treatment (e.g., immobilization, oral NSAIDs, local corticosteroid injections) for more than 3 months;
6. Signing the informed consent form.

Exclusion Criteria:

1. Ultrasound examination reveals bifurcation of the median nerve or the presence of a persistent median artery at the carpal tunnel entrance, or compression at the carpal tunnel caused by cysts, tumors, or fracture fragments;
2. Systemic infection or local infection at the surgical site;
3. Severe coagulation disorders;
4. Previous carpal tunnel syndrome surgery on the affected side for this operation;
5. Patients with uncontrolled epilepsy, cervical radiculopathy, or diabetic peripheral neuropathy;
6. Allergy to local anesthetics;
7. Inability to complete the questionnaire due to language or cognitive impairments;
8. Patients with severe heart, lung, liver, or brain diseases;
9. Patients with mental illnesses;
10. Participation in other clinical trials within the last three months;
11. Pregnant or breastfeeding women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in BCTQ scale scores compared to preoperative values at 6 months postoperatively | 6 months post-operation
  The Boston Carpal Tunnel Questionnaire (BCTQ) is considered an effective tool for assessing the severity of symptoms and functional status in carpal tunnel syndrome. It is divided into two parts: the Symptom Severity Scale (SSS) and the Functional Status Scale (FSS). The SSS consists of 11 questions that evaluate the severity, frequency, and duration of symptoms. The FSS comprises 8 questions that assess the impact of the syndrome on daily life activities. Each question is scored from 0 (no symptoms or no impact) to 5 (most severe). The total score of the questionnaire is the average score of all questions.

SECONDARY OUTCOMES:
quickDASH scale score | preoperative, 2 weeks, 3 months, and 6 months postoperative
  The change in Quick Disabilities of the Arm, Shoulder and Hand (quickDASH) scores from preoperative to 2 weeks, 3 months, and 6 months postoperative. Researchers will ask the enrolled patients the questionnaire either in person, over the phone, or online, then record the answers, summarize, and document the scores.
Grip strength | before the surgery, 6 months postoperative
  The change in grip strength from before the surgery to 6 months postoperative. Researchers will explain the use of the dynamometer to the patients, assist them in measuring their grip strength, and record the dynamometer readings.
Pinch strength | before the surgery, 6 months postoperative
  The change in pinch strength from before the surgery to 6 months postoperative. Researchers will explain the use of the dynamometer to the patients, assist them in measuring their pinch strength, and record the dynamometer readings.
the cross-sectional area of the median nerve at the proximal entrance of the carpal tunnel under ultrasound | before the surgery, 6 months postoperative
  The comparison of the cross-sectional area of the median nerve at the proximal entrance of the carpal tunnel under ultrasound between preoperative and 6 months postoperative. This will be examined and reported by the Ultrasound Department of our hospital.
Time to return to work | 1, 2, and 4 weeks postoperative
  The time to return to work after surgery is defined as the number of days from the day of surgery to the first day the patient returns to their preoperative job or is able to fully resume daily activities. This is self-assessed by the patient, and researchers will ask and record the information at 1, 2, and 4 weeks postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China